CLINICAL TRIAL: NCT06677554
Title: COVARIAN - Contribution of Contrast Enhanced Ultrasound for Diagnosis of Adnexal Torsion: a Randomized Controlled Trial
Brief Title: Contribution of Contrast Enhanced Ultrasound for Diagnosis of Adnexal Torsion
Acronym: COVARIAN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BERTHOLDT Charline, Clinical Professor, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021PI162
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Adnexal Torsion
MeSH Terms: conditions — Ovarian Torsion | interventions — Contrast Media; contrast agent BR1; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound with contrast injection (Experimental): Patients consulting the gynecological emergencies as part of the management of a strong suspicion of adnexal torsion (after the clinical examination and standard ultrasound)
  Interventions: Drug: Addition of ultrasound with contrast injection (SonoVue®)
- Control (Active Comparator): Patients consulting the gynecological emergencies as part of the management of a strong suspicion of adnexal torsion (after the clinical examination and standard ultrasound)
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Drug: Addition of ultrasound with contrast injection (SonoVue®) — Addition of contrast evaluation with SonoVue® injection (5 min including 1 min of acquisition) within the diagnostic strategy
  Arms: ultrasound with contrast injection
Other: Standard Care (in control arm) — No addition of ultrasound with contrast
  Arms: Control

SUMMARY:
Adnexal torsion is the rotation of the ovary around its vascular axis resulting, in the absence of treatment, ischemia that can lead to peritonitis by necrosis or impaired fertility. It is a gynecological emergency affecting 3% of women of childbearing age, including from adolescence, and requires surgical treatment as soon as possible, classically within 6 hours.

The symptomatology of adnexal torsion is dominated by pelvic pain of sudden onset and variable intensity, an aspecific sign that does not allow a diagnosis of certainty. There are no biological markers and, in the context of the emergency, the only imaging examination available is pelvic ultrasound associated with a Doppler flow analysis but with a low and variable diagnostic performance depending on the studies (sensitivity variable from 46 to 73%).

There are currently no tests that can provide a diagnosis of certainty. Only surgical exploration, carried out at the discretion of the practitioner on the basis of a bundle of arguments, can confirm or refute the diagnosis. However, this management strategy leads to the realization of emergency surgical interventions wrongly since 3 out of 10 women will finally not have an adnexal torsion (PMSI data from participating centers: 30 to 45% false positives).

Contrast ultrasound is a technique that uses a strict intravascular product to assess the vascularization of the ovary and offers a high diagnostic performance in the context of adnexal torsion. Indeed, a retrospective study, published in 2021, reports a sensitivity of 94% and a specificity of 100%. The preliminary results of our pilot study (AGATA APJC 2019, Dr Bertholdt, NCT04522219) also go in this direction with a sensitivity of 100%, a specificity of 86% and a negative predictive value of 100% (data being published).

The COVARIAN project, second stage of the AGATA project, aims to demonstrate that the addition of a contrast evaluation to standard ultrasound in the diagnostic strategy in case of suspicion of adnexal torsion improves the health of women by reducing the rate of wrongly surgery, that is, without proven torsion.

COVARIAN will be the first prospective multicenter randomized study evaluating the direct benefit for women of using ultrasound contrast evaluation in the management strategy in case of suspicion of adnexal torsion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or over
* Person who has carried out a preliminary clinical examination adapted to the clinical trial
* Strong suspicion of adnexal torsion with surgery planned
* No ongoing pregnancy or breastfeeding
* Affiliation to or beneficiary of a social security scheme
* Person who has received complete information on the organization of the research and has signed their informed consent

Exclusion Criteria:

* Person who does not understand and/or speak French
* Any medical situation that does not indicate the administration of SonoVue®, including:

  * Known hypersensitivity to sulphur hexafluoride or any of the other components of SonoVue
  * Woman with acute coronary syndrome or unstable ischemic heart disease
  * Woman with acute endocarditis
  * Woman with valve prostheses
  * Women with acute systemic inflammatory disease and/or sepsis
  * Woman with hypercoagulation and/or recent thromboembolic accident
  * End-stage woman with kidney or liver disease
  * Woman with right-left shunt, severe pulmonary hypertension (pulmonary arterial pressure > 90 mmHg)
  * Women with uncontrolled systemic hypertension
  * Woman with respiratory distress syndrome
  * Medical condition contraindicating the administration of SonoVue®,
* History of PEG allergy (or macrogol)
* Person referred to in Articles 10, 31, 32, 33 and 34 of Regulation EU 536/2014:

  * Pregnant, parturient or breastfeeding/nursing mother
  * Minor (not emancipated)
  * Adult subject to a legal protection measure (guardianship, curatorship, safeguarding of justice)
  * Person of legal age who is unable to express consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 256 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2028-02-07 (Estimated); Study Completion 2028-02-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the two-stage diagnostic strategy effectiveness | 38 months
  Percentage of surgical procedures performed in emergency (within 6 hours of arrival of the patient) without proven torsion (no visible spiral turn in intraoperative) in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Charline BERTHOLDT, Pr, Principal Investigator — CHRU Nancy
Locations (6):
- France (6):
  - CHU, Besançon
  - CHU, Dijon
  - CHRU Nancy - Maternité Régionale, Nancy
  - CHU, Reims
  - CMCO, Schiltigheim
  - CHU Hautepierre, Strasbourg

IPD SHARING:
Plan to Share IPD: No